CLINICAL TRIAL: NCT06076538
Title: Prospective Observational Study Using PET/MR for Characterization of Renal Masses (RMs)
Brief Title: PET/MR for Characterization of Renal Masses (RMs)
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Principal Investigator, Robert Sibley, Assistant Professor, Radiology, University of Texas Southwestern Medical Center
Other Study IDs: STU-2022-1158
Record Dates: First submitted 2023-09-06; First posted 2023-10-11 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Renal Tumor; Renal Cell Carcinoma; Renal Tumor, Benign
Keywords: Renal Mass; Renal Cell Carcinoma; PET/MR
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For patients undergoing standard of care biopsy, an extra core will be obtained for future research from participants who opt-in to have extra core collected when they sign informed consent form. If the renal mass is resected surgically, a piece of discarded tissue will be collected for similar correlative studies. The extra core or the discarded tissue will be used for metabolomics analysis to understand the correlation of FDG uptake and tumor metabolism.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient diagnosed with incidental solid renal mass: All patients at our institution who are diagnosed with indeterminate solid SRM and without prior treatment for the tumor, renal biopsy or contraindication to PET/MRI can be included in the study. This will be a prospective, non-randomized, non-blinded observational study. Patients will then be managed following the standard of care.
  Interventions: Diagnostic Test: 2-Deoxy-2-[18F]fluoroglucose Positron Emission Tomography/Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: 2-Deoxy-2-[18F]fluoroglucose Positron Emission Tomography/Magnetic Resonance Imaging — PET/MR scan utilizing FDG Radiopharmaceutical
  Other Names: FDG PET/MR

SUMMARY:
The frequency of kidney tumors found incidentally on imaging studies performed for unrelated reasons continues to increase leading to more surgeries and ablations for the treatment of renal masses thought to be cancer. However, about 20% of these masses are not cancerous and do not require treatment. Many cancerous kidney tumors are indolent and can be followed safely with imaging (i.e., particularly tumors <2 cm and in patients with limited life expectancy), while some tumors are both malignant and aggressive, with a higher potential to spread outside the kidney and require treatment.

The purpose of this observational study is to assess the ability of Fludeoxyglucose (18F) (FDG) PET/MR to distinguish different types of kidney tumors. The investigators hypothesize that PET/MR will better show differences between aggressive and both indolent and benign kidney masses compared to the currently used radiologic scans.

Participants will be selected from those who have been scheduled to receive a contrast-enhanced MRI for their regular care due to a suspicious kidney mass. Participants will have their MRI on a hybrid PET/MR scanner capable of obtaining both MRI and PET images. While they are receiving their standard of care MRI exam, patients will also receive a research FDG PET exam. Participants will have an IV placed for administration of the MRI contrast agent, just as they would if they were not taking part in the study. The same IV will be used to give the FDG radiopharmaceutical for the PET scan and furosemide (a diuretic), to help empty the bladder before the scan and help better see the kidneys on the scans. Both FDG and furosemide are FDA approved medications. Participants will have only one visit with the research team which will last ~2.5 hours and will include collection of the participant's regularly scheduled MRI.

If participants undergo surgery to remove the tumor, the study will collect samples of the removed tissue for research. If participants receive a biopsy of the tumor, the study may collect an additional sample of the tumor for research.

After the PET/MRI, participants will not have additional visits with the study team, but the study team may call every 6-12 months for up to 2 years to see how they are doing and ask about their health. The study team will review the medical record for any changes to their diagnosis, updates to their medical history, new scans ordered by their regular doctor, or recent lab or biopsy results.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is most commonly diagnosed as an incidental small renal mass (SRM, ≤4cm [cT1a]). The incidence of RCC has markedly increased in the last few decades due to the widespread utilization of cross-sectional imaging. The increased detection of renal masses has resulted in an accompanying increase in the number of surgeries and ablations performed for a mass suspected of being a cancer. However, despite aggressive treatment of SRMs over the last few decades, there has not been a substantial decrease in kidney cancer-specific mortality suggesting an over-treatment effect - i.e., many patients may not benefit from extirpative or ablative treatment. Furthermore, approximately 20% of small (≤4 cm) solid renal masses are benign neoplasms, mostly oncocytoma and angiomyolipoma. Benign masses generally do no harm and can be ignored or followed up as they do not limit a patient's lifespan. Even when malignant, small solid masses are frequently indolent with low rates of local disease progression or metastasis. The proportion of benign diagnoses and indolent RCCs is higher among solid masses smaller than 2 cm. Although percutaneous renal mass biopsy can offer a definitive diagnosis, it is not feasible in every patient, and carries a high non-diagnostic rate (14-19%), has low negative predictive value (63%) and underestimates tumor grade. For these reasons, combined with a desire to identify aggressive renal masses with increased risk of progression or metastasis promptly and decrease patient morbidity and health-care costs related to unnecessary treatments, there is a need for developing imaging techniques that better characterize renal masses. In addition to differentiating benign from malignant disease, distinction between indolent malignant renal masses from aggressive neoplasms is important for decision making, with the later typically requiring prompt intervention. In contrast, active surveillance may be favored for patients with indolent malignancies, particularly for those with competing comorbidities and limited life expectancy. Unfortunately, the lack of reliable predictors of oncologic behavior have also limited the wide clinical adoption of active surveillance as a management strategy. Aggressive renal masses are classified by the presence of any high grade (HG, International Society of Urogenital Pathology (ISUP) grade 3 or 4 out of 4) features on histology or the presence of sarcomatoid and rhabdoid features, coagulative necrosis.

Alternatively, a diagnosis of the histologic subtype of RCC may assist in management decisions. For example, clear cell renal cell carcinoma (ccRCC) is the most common histology and metastasizing tumor. The clear cell likelihood score (ccLS) is a 5-tier system developed at the University of Texas Southwestern Medical Center (UTSW) to predict the likelihood of a solid renal mass to represent a clear cell renal cell carcinoma. In a multicenter, retrospective study, the reported pooled sensitivity, specificity, and positive predictive value for ccRCCs using a ccLS of 4 or 5 were 75% (95% CI: 68, 81), 78% (95% CI: 72, 84), and 76% (95 CI: 69, 81), respectively. The negative predictive value for a ccLS of 1 or 2 was 88% (95% CI: 81,93).

Patients referred for MRI of an indeterminate renal mass will be eligible for this study. PET/MRI in this study will be performed as a replacement of the standard-of-care MRI examination. Thus, the PET component of the PET/MR examination is a research procedure. Patients will be screened for any contraindication of MRI (e.g., unsafe indwelling device) as it is routinely done in the Department of Radiology for clinical MRI examinations. Patients will be administered with 12 mCi of FDG I.V, which is consistent with the FDG radiation dose patients receive for FDG PET/CT examinations performed as standard of care. Patients will receive 20 mg of furosemide 60 min after administration of FDG. The patient will be asked to empty their bladder as much as needed for the following 60 min. The patient will then be placed on the PET/MRI table 60 min after administration of FDG for a 10 min quick PET/MR acquisition the abdomen. The patient will be removed from the scanner and asked to empty their bladder as needed. The patient will be placed on the MRI scanner again 120 min after the administration of FDG to complete their standard of care MRI. A gadolinium-enhanced MRI of the kidneys will be obtained using the standard clinical protocol for MRI of renal masses at UTSW. An extracellular gadolinium-based contrast agent will be administered during the MRI and is not part of the study procedures. PET data of the kidneys will be acquired simultaneously during the MRI examination as part of the study procedures. UTSW standard operating procedures will be followed with regards to fasting and blood glucose measurements for patients undergoing FDG PET imaging in this study. PET images will be coregistered to MRI data and mean and maximum standardized uptake value in the renal mass will be calculated. MRI images will be interpreted using the standard clinical report and a ccLS will be provided. For patients undergoing standard of care biopsy, an extra core will be obtained for future research from participants who opt-in to have extra core collected when they sign informed consent form. If the renal mass is resected surgically, a piece of discarded tissue will be collected for similar correlative studies. The extra core or the discarded tissue will be used for histology and metabolomics analysis to understand the correlation of FDG uptake and tumor metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known solid (>25% total volume enhances) renal mass
* Renal mass size measuring >2 to ≤7 cm
* Age >18 years
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Pregnancy
* Prior percutaneous biopsy of the renal mass
* Prior treatment of the renal mass
* Prior hemorrhage in the renal mass
* Contraindication to MRI or PET
* Renal mass not eligible for ccLS based on prior imaging (i.e., containing macroscopic fat [classic angiomyolipoma] or enhancing less than 25% of its volume [considered a cystic renal mass])
* Genetic syndrome predisposing to renal masses (e.g., VHL, BHD, TSC, etc.);
* More than 3 renal masses at time of initial diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will complete their clinically indicated MRI with the addition of the research infusion of the FDA approved FDG radiotracer and PET portion of the scan. Eligibility waivers are not permitted. Subjects must meet all of the inclusion and exclusion criteria to be registered to the study.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of SRM aggressiveness with PET | Baseline
  To test the difference in mean SUVmax between HG malignant renal masses and other (LG malignancies and benign) renal masses.

SECONDARY OUTCOMES:
Prediction of SRM aggressiveness with the metabolic clear cell likelihood score (m-ccLS) | Baseline
  To determine the diagnostic performance of combining SUVmax and clear cell likelihood score (ccLS; ranging from 1 (very unlikely) to 5 (very likely)) in detecting HG SRM size >2 to ≤7 cm and compare to that of ccLS alone.
Prediction of aggressive clear cell histology with the metabolic clear cell likelihood score (m-ccLS) | Baseline
  To determine the diagnostic performance of combining SUVmax and clear cell likelihood score (ccLS; ranging from 1 (very unlikely) to 5 (very likely)) in detecting HG ccRCC from all solid SRM size >2 to ≤7 cm and compare to that of ccLS alone.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Pedrosa, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared.